CLINICAL TRIAL: NCT06314737
Title: Assessment of Efficacy of New Adjuvant Therapy in Locally Advanced Rectal Cancer
Brief Title: Assessment of Efficacy of Neoadjuvant Therapy in Locally Advanced Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Cai Zerong, Deputy Chief Physician, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: 2021ZSLYEC-192
Record Dates: First submitted 2024-03-09; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Locally Advanced Rectal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The pathological specimens before operation and the specimens after operation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neoadjuvant therapy group: The primary tumor received neoadjuvant therapy before surgical treatment.
- Surgical treatment group: The primary tumor did not receive neoadjuvant therapy before surgical treatment.

SUMMARY:
This study analyzed the efficacy differences between neoadjuvant therapy and direct surgical treatment in patients with locally advanced rectal cancer in the real world. The aim was to evaluate the impact of neoadjuvant therapy on overall survival, disease-free survival, and local recurrence-free survival in patients with locally advanced rectal cancer, explore the population benefiting most from neoadjuvant therapy, and provide evidence-based medicine for the benefits of neoadjuvant therapy in patients with colorectal cancer in the real world.

DETAILED DESCRIPTION:
Colorectal cancer ranks third in terms of global incidence (10.2%) and second in terms of mortality (9.2%) among malignant tumors, with rectal cancer accounting for one-third of cases. The standard treatment regimen for locally advanced rectal cancer (LARC), neoadjuvant chemotherapy (NACT) combined with total mesorectal excision (TME), has been shown to better control local disease, reduce local recurrence rates, but does not improve overall survival. In recent years, with the continuous improvement of surgical techniques, surgical treatment has also achieved better local control effects for locally advanced rectal cancer. However, the efficacy of neoadjuvant therapy varies greatly in different studies. For locally advanced rectal cancer, a prospective clinical study published in the New England Journal of Medicine in 2004 compared the efficacy differences between preoperative neoadjuvant chemoradiotherapy (NCRT) and postoperative chemoradiotherapy. The study demonstrated that compared to postoperative chemoradiotherapy, preoperative NCRT combined with total mesorectal excision could better control the local disease, reduce the toxicity of chemoradiotherapy, but did not help prolong overall survival. However, due to issues such as increased postoperative complications associated with neoadjuvant radiotherapy, some rectal cancer patients refuse neoadjuvant radiotherapy. Therefore, a significant amount of research has also been devoted to proving the efficacy of neoadjuvant chemotherapy alone.

Additionally, neoadjuvant therapy can also increase the rate of sphincter preservation for low rectal cancer. However, there is still controversy over whether neoadjuvant therapy can bring survival benefits to rectal cancer patients. How to reduce overtreatment caused by neoadjuvant therapy and related toxic side effects is also a current research hotspot. This study analyzed the efficacy differences between neoadjuvant therapy and direct surgical treatment in patients with locally high-risk rectal cancer in the real world, aiming to evaluate the impact of neoadjuvant therapy on overall survival, disease-free survival, and local recurrence-free survival in patients with locally high-risk rectal cancer, explore the high-benefit population of neoadjuvant therapy, and provide evidence-based medicine evidence for the benefits of neoadjuvant therapy in real-world rectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological examination confirmed primary rectal adenocarcinoma;
2. Pelvic MRI or abdominal-pelvic CT at initial diagnosis diagnosed as T3-4 or N+;
3. Thoracoabdominal CT indicated no evidence of distant metastasis;
4. Distance from the tumor lower margin to the anal verge ≤12cm;
5. Underwent surgical treatment.

Exclusion Criteria:

1. Concurrently diagnosed with multiple colorectal cancers or concomitant other malignant tumors;
2. Locally recurrent rectal cancer;
3. Initial diagnosis suggests suspicious distant metastasis;
4. Histological diagnosis of rectal squamous cell carcinoma, adenocarcinoma, or neuroendocrine carcinoma;
5. MRI information lost;
6. Did not undergo surgical treatment;
7. Upper rectal cancer or cancer at the rectosigmoid junction.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who visited the Sixth Affiliated Hospital of Sun Yat-sen University between October 2010 and December 2018, were diagnosed with primary rectal adenocarcinoma based on initial pathological examination, and were diagnosed as T3-4 or N+ based on pelvic MRI or abdominal-pelvic CT scan. Their distance from the tumor lower margin to the anal verge was ≤12cm, and they subsequently underwent surgical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 3515 (Actual)
Dates: Start 2010-10-02 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival | From date of randomization until the date of death from any cause, assessed up to 120 months
  Overall survival is defined as the time from the date of randomization to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Zerong Cai, MD, Study Director — Sixth Affiliated Hospital, Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No
Please contact us by e-mail

REFERENCES:
- [Derived] Wang Z, Bai F, Chen Y, Liu X, Huang Z, Zhu Q, Wu X, Cai Z. Does the initial treatment of primary tumor impact prognosis after recurrence in locally advanced rectal cancer? Results from a retrospective cohort analysis. Int J Colorectal Dis. 2024 Sep 28;39(1):153. doi: 10.1007/s00384-024-04721-9. PMID 39333450